CLINICAL TRIAL: NCT05633394
Title: Subcostal Temporary Extravascular Pacing V (STEP V) Study
Brief Title: Subcostal Temporary Extravascular Pacing V Study
Acronym: STEP V
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AtaCor Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: DOC-10235
Record Dates: First submitted 2022-11-22; First posted 2022-12-01 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Conduction Defect
Keywords: Temporary Ventricular Pacing; Extravascular
MeSH Terms: conditions — Arrhythmias, Cardiac

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AtaCor EV Temporary Pacing Lead System (Experimental): Subjects implanted with the AtaCor StealthTrac Lead Model AC-101400
  Interventions: Device: AtaCor StealthTrac Lead

INTERVENTIONS:
Device: AtaCor StealthTrac Lead — Subjects will receive the AtaCor StealthTrac Lead being evaluated in the study.

SUMMARY:
The STEP V Study is a prospective, multicenter, acute (in-hospital), single-arm feasibility study. The objective of the study is to evaluate the early safety and performance of the latest AtaCor EV Temporary Pacing Lead System over a two-day use period.

DETAILED DESCRIPTION:
The primary safety objective is freedom from Adverse Device Effects (ADE). The primary performance objective is summary statistics for pacing capture threshold, impedance, and sensed R-wave amplitude with the StealthTrac Lead from insertion through removal.

Up to three (3) Investigational Sites will participate with up to 50 subjects enrolled in the study. Subjects indicated for closed-chest cardiac invasive procedures will be eligible for participation. Subjects undergoing a qualifying index procedure will have a Model AC-101400 StealthTrac Lead inserted and evaluated over the follow-up period. Subject participation is expected to be 2 days with the Study Lead inserted, plus 30 days post lead removal. A 30 day (+/-3 days) post-removal follow-up will also be performed to document any latent adverse events. Subjects remain enrolled until completion of the 30-Day Follow Up.

The maximum duration for study participation is 33 days. Study duration estimated to be 3 years after the first study enrollment.

ELIGIBILITY:
Inclusion criteria

1. At least 18 years old
2. Subjects indicated for closed-chest cardiac invasive procedure, including:

   * Transarterial transcatheter aortic valve implantation (TAVI)
   * Transarterial balloon aortic valvuloplasty (BAV)
   * Cardiovascular implantable electronic device (CIED) pulse generator replacement
   * Cardiovascular implantable electronic device (CIED) lead extraction or revision

Exclusion criteria

1. BMI ≥ 35 kg/m2
2. Septic shock
3. Severe anemia
4. Patients on dual antiplatelet therapy or anti-coagulation that cannot be stopped for the procedure
5. Circumstances that prevent data collection or follow-up (e.g., inability to perform a short walk with the Holter monitor)
6. Participation in any concurrent clinical study without prior written approval from the Sponsor
7. Inability or unwillingness to provide informed consent to participate in the Study

   Known prior history for any of the following:
8. Median or partial sternotomy
9. Acute coronary syndrome within past 90 days
10. NYHA Functional Classification IV within past 90 days
11. Surgically corrected congenital heart disease (not including catheter-based procedures)
12. Allergies to the device materials such as stainless steel, titanium, platinum, iridium, polyethylene, polyurethane, polycarbonate and silicone
13. Surgery with disruption of the lung, pericardium or connective tissue between the sternum and pericardium, including adhesions
14. Significant anatomic derangement of or within the thorax (e.g., pectus excavatum, significant scoliosis)
15. Thoracic radiation therapy, pneumothorax, pneumomediastinum or other medical treatments which may complicate the AtaCor EV Temporary Pacing Lead System insertion procedure
16. Any conditions which may complicate the AtaCor EV Temporary Pacing Lead System insertion procedure
17. Pericardial disease, pericarditis and mediastinitis
18. Medical treatments, surgeries or conditions that increase the potential for pericardial adhesions
19. FEV1 < 1 liter

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2023-01-23 (Actual); Primary Completion 2025-05-29 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Freedom from ADEs | Up to 2 days post-insertion
  Freedom from Adverse Device Effects (ADE)
Pacing Capture Threshold (mA or V) | Up to 2 days post-insertion
  Summary statistics for pacing capture threshold with the StealthTrac Lead from insertion through removal
Impedance (Ohms) | Up to 2 days post-insertion
  Summary statistics for impedance with the StealthTrac Lead from insertion through removal
Sensed R-Wave Amplitude (mV) | Up to 2 days post-insertion
  Summary statistics for sensed R-wave amplitude with the StealthTrac Lead from insertion through removal

CONTACTS AND LOCATIONS:
Overall Officials: Martin C Burke, DO, Principal Investigator — AtaCor Medical, Inc.
Locations (1):
- Sanatorio Italiano, Asunción, Paraguay